CLINICAL TRIAL: NCT04848818
Title: Multicenter Prospective Trial for Operative Treatment of Distal Pediatric Forearm Fractures With PLGA-based Biodegradable Material (Activa Im-Nails™) and Conventional Implants (K-wires)
Brief Title: Comparative Trial of Operative Treatment of Distal Pediatric Forearm Fractures With Biodegradable Nails and K-wires
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Péterfy Sándor Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 228-01-CIP-3
Record Dates: First submitted 2021-04-08; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-03

CONDITIONS: Fracture Wrist
Keywords: children; radius; fracture; wire; bioabsorbable
MeSH Terms: conditions — Wrist Fractures; Fractures, Bone | interventions — Drug Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- K-wire group (Active Comparator): Children with closed or grade I. open, severly displaced distal radial and/or complete forearm metaphyseal fractures between the age 3-13.
  Interventions: Procedure: Distal radial metaphyseal fracture fixation with percutaneous K-wires
- Activa-IM Nail group (Active Comparator): Children with closed or grade I. open, severly displaced distal radial and/or complete forearm metaphyseal fractures between the age 3-13.
  Interventions: Procedure: Distal radial and/or ulnar metaphyseal fracture fixation with bidegradable PLGA-based (Activa Im-Nail) implants

INTERVENTIONS:
Procedure: Distal radial metaphyseal fracture fixation with percutaneous K-wires — Pediatric distal metaphyseal fractures which are severly displaced will be operated with percutaneous K-wires..
  Arms: K-wire group
Procedure: Distal radial and/or ulnar metaphyseal fracture fixation with bidegradable PLGA-based (Activa Im-Nail) implants — Pediatric distal metaphyseal radial and /or ulnar fractures which are severly displaced will be operated with percutaneous bidegradable PLGA-based (Activa Im-Nail) implants.
  Arms: Activa-IM Nail group

SUMMARY:
The study is designed as a multicenter trial for the treatment of distal pediatric forearm fractures (=severely displaced distal metaphyseal forearm fractures) with a PLGA-based biodegradable intramedullary implant in children. The primary objective of the trial is to evaluate clinical outcome between Activa IM-Nail™ and K-wire in this indication. The secondary objective is to evaluate potential differences of potential complications in the operative method with either a biodegradable intramedullary PLGA-implant or with conventional K-wires. K-wire osteosynthesis will be made according to the conventional surgical technique by three paediatric trauma centers. Intramedullary PLGA implantation will be made by the Péterfy Hospital. The surgical indication will be the same in all groups, and follow-up will follow standard protocols. In the further clinical course, the patients in the study group treated with PLGA implants spare a subsequent operation for implant removal after 4-8 weeks. The results of different surgeries will be compared based on several criteria.

DETAILED DESCRIPTION:
Over the last decade, there has been an increasing demand to overcome the disadvantages associated with conventional implant materials, by developing new, alternative materials and material production approaches for use in trauma care.

In recent years there has been a growing interest in the orthopaedic application of resorbable implants. Their use in children may be particularly beneficial. Poly(L-lactide)-co-glycolide acid (PLGA) is a well-known, reliable biodegradable material that has been used in bone surgery for more than 20 years. Several publications have already reported the successful use of intra-medullar PLGA implants in the treatment of paediatric diaphyseal forearm fractures.

To gather further evidence about the clinical value of the new method with PLGA - based bioresorbable implant in regard to patients benefit, a multicenter prospective trial is needed. This trial will be conducted on the distal forearm, which is one of the most common fracture locations that requires surgical intervention in children. Severely displaced distal paediatric forearm fractures will be addressed.

Distal paediatric forearm injuries

Distal radius fractures are among the most common injuries of childhood. Optimal treatment for distal radius fractures is still controversial. Treatment of severely displaced and shortened fractures usually require general narcosis and closed reduction. Most authors recommend osteosynthesis if the fracture remains unstable after reduction. The gold standard operative method for these fractures is closed reduction, percutaneous pinning with Kirschner-wires.

Kirschner-wire related minor complications are relatively frequent. Migration of the pins, superficial infections, skin irritation are well manageable but significantly impair the child's sense of comfort. Deep infections, tendon or nerve injuries may occur less often. There is a controversy as to whether it is preferable to leave the wires outside the skin. While wires left out of the skin increase the risk of infection, wires buried under the skin can be removed with a second intervention. Removing the implants can also cause complications.

K-wires are not capable of providing sufficient stabilization in this indication, so additional casting treatment is also required. The duration and the type of postoperative immobilization varies greatly according to the practice of the surgeons. There is no evidence about the most optimal immobilization procedure. 4-6 weeks of cast wearing is recommended by most authors. This causes stiffness in the affected joints and delays the recovery of full function. Fractures with intramedullary elastic nails require a reduced time of immobilization because they provide a more stable synthesis, but nails can be removed only under general anaesthesia. The use of bioabsorbable intramedullary nails in distal paediatric forearm fractures may eliminate all of the above-mentioned disadvantages.

The study is designed as a multicenter trial for the treatment of distal pediatric forearm fractures (=severely displaced distal metaphyseal forearm fractures) with a PLGA-based biodegradable intramedullary implant in children. The primary objective of the trial is to evaluate clinical outcome between Activa IM-Nail™ and K-wire in this indication. The secondary objective is to evaluate potential differences of potential complications in the operative method with either a biodegradable intramedullary PLGA-implant or with conventional K-wires. K-wire osteosynthesis will be made according to the conventional surgical technique by two paediatric trauma centers. Intramedullary PLGA implantation will be made by the Péterfy Hospital. The surgical indication will be the same in all groups, and follow-up will follow standard protocols. In the further clinical course, the patients in the study group treated with PLGA implants spare a subsequent operation for implant removal after 4-8 weeks. The results of different surgeries will be compared based on several criteria.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of distal radial or complete forearm fracture Metaphyseal radial/or distal forearm fractures with complete displacement and shortening.

Age between of 3-13 years. Open physeal plates on X-rays. Closed or Grade I. open fractures Ability and willingness to give an informed consent

Exclusion Criteria:

Pathological fractures (e.g. bone cyst) Poly-traumatized patient Inability or unwillingness to give informed consent Closed physeal plates on X-rays. Active skin infection in the surgical area

Ages: 3 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 164 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Does the short intramedullary nailing operative method with bioabsorbable Activa IM Nails™ correlate to less complications than the conventional K- wiring technique in displaced pediatric distal forearm or radial metaphyseal fractures? | Six months after operation
  We compare the incidence of minor and major complications of both surgical technique. These are: superficial skin infection, tendon injury, nerve injury, secondary displacement, deep infection, skin irritation.

SECONDARY OUTCOMES:
Does the short intramedullary nailing operative method with bioabsorbable Activa IM Nails™ also reduce the postoperative immobilisation time? | Eight weeks after operation
  Calculation of postoperative immobilisation time in weeks. Calculation and comparison the necessary immobilisation times in both surgical techniques.
Does the short intramedullary nailing operative method with bioabsorbable Activa IM Nails™ not require a second intervention? | Six months after operation
  Calculation and comparioson of the number of a second operative intervention in both surgical techniqes.
Does the short intramedullary nailing operative method with bioabsorbable Activa IM Nails™ also reduce the postoperative outpatient visits? | 1 year after operation
  Calculation and comparison the number of postoperative outpatient visits in both surgical techniques.
Does the short intramedullary nailing operative method with biodegradable nails and K-wire technique results a full recovery of the functions within six months? | Six months after operation
  Examination by the range of motion method (ROM) of the wrists of the patients. Full recovery means , that the range of pronation/supination and flexion/extension of the wrist will be the same as the range of the healthy side.The examination is also performed at weeks 4,8,and 24.
Does the short intramedullary nailing operative method with biodegradable nails shortens the recovery time for the full function compared to the K-wiring method? | Six months after surgey
  Based on the results of ROM -method examinations performed at weeks 4,8 and 24 weeks ,we compare and calculate the difference in the rates of function recovery in both surgical technique.

CONTACTS AND LOCATIONS:
Overall Officials: Marcell Varga, PhD, Principal Investigator — Péterfy Hospital, National Trauma Center,Budapest
Locations (4):
- Hungary (4):
  - Szent János Hospital, Budapest, Diós Árok 1.
  - Péterfy Hospital, Budapest, Fiumei Út 17
  - Medical University of Pécs, Pediatric Surgery, Pécs, József Attila U 7.
  - Heim Pál Hospital, Budapest, Üllöi Út 86

IPD SHARING:
Plan to Share IPD: No